CLINICAL TRIAL: NCT00967096
Title: Rifaximin for Preventing Acute Graft Versus Host Disease
Brief Title: Rifaximin for Preventing Acute Graft Versus Host Disease (AGVHD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, John Horan, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00003578; Rifaximin (Other: Other)
Record Dates: First submitted 2009-08-11; First posted 2009-08-27 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Malignancy; Bone Marrow Transplantation
Keywords: rifaximin; acute graft versus host disease; bone marrow transplant; non-malignancy requiring BMT
MeSH Terms: conditions — Neoplasms | interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): The primary clinical endpoint to be assessed in this study will be the proportion of Rifaximin doses successfully administered. Because of mucositis, compliance with oral agents, even those that are well tolerated in other settings, may be limited in the early post-transplant period. Thus, it will be important to demonstrate the feasibility of administering Rifaximin to BMT patients before embarking on larger scale studies. Secondary outcomes will include AGVHD, event-free survival, overall survival, non-relapse mortality, neutrophil and platelet engraftment.
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: Rifaximin — Rifaximin for Bone marrow transplant patients

SUMMARY:
Acute graft versus host disease is a frequent and often life threatening complication of allogeneic blood and marrow transplantation. The bacteria that normally reside in the intestine play a critical role in its development. Injury to the lining of the bowel that results from the high dose chemotherapy or radiation that transplant patients receive during the week preceding the transplant allows the bacteria to invade the intestines and spread to nearby lymph nodes. This, in turn, causes inflammation which has been shown to promote GVHD. Both pre-clinical and clinical research has demonstrated that oral antibiotics can prevent graft versus host disease by inhibiting these gut bacteria. Rifaximin has several features that suggest it could be effective in preventing GVHD. Rifaximin prophylaxis might also provide an added benefit by protecting highly immunocompromised transplant patients from severe bacterial infections. This pilot trial will allow the investigators to determine the feasibility of using Rifaximin for prevention of GVHD and infection in patients undergoing allogeneic blood and marrow transplantation. The preliminary results will be used to plan a more definitive trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be at least 12 years old.
2. Patients will be eligible regardless of their type of disease (malignant or non-malignant), type of donor (HLA matched related, mismatched related or unrelated donors), type of hematopoietic cell source (unstimulated marrow, cytokine stimulated marrow, cytokine stimulated peripheral blood or umbilical cord blood), or GVHD prophylaxis.
3. Patients must receive a myeloablative or moderately intensive reduced intensity (at least 8 mg/kg oral busulfan (or the equivalent IV dose), or at least 100 mg/m2 of Melphalan , or at least 100 mg/kg of cyclophosphamide, or at least 500 cGy of TBI) conditioning regimen.

Exclusion Criteria:

1. Age under 12 years.
2. Known hypersensitivity to rifaximin, or other rifamycin antimicrobial agents.
3. Minimally toxic conditioning regimen (e.g. low dose TBI based). Since these regimens induce minimal myelosuppression and gut injury, patients receiving them probably stand little to gain from antibiotic prophylaxis.
4. Patients with documented severe active infection (viral, bacterial, fungal, protozoal) will not be eligible.
5. Patients with treatment unresponsive hematologic malignant diseases (based on an assessment done within two weeks of the start of conditioning therapy).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Determine the feasibility of this approach; to gather preliminary data on the incidence of GVHD and other clinical outcomes; to obtain pre-clinical data on the serial plasma levels of three biologic markers- endotoxin, soluble IL-2 receptor and TNF. | 1 year after last patient enrolled

SECONDARY OUTCOMES:
Obtain preliminary data on the efficacy of administering rifaximin for prophylaxis against serious bacterial infections in BMT patients. | 1 year after last patient enrolled

CONTACTS AND LOCATIONS:
Overall Officials: John Horan, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Emory University, Atlanta, Georgia